CLINICAL TRIAL: NCT03037801
Title: Prospective Randomized Controlled Study of the Use of Intrapulmonary Percussive Ventilation (IPV) for Children With Bronchiolitis Admitted to the Pediatric Intensive Care Unit (PICU) and Are on Non-Invasive Ventilation Support
Brief Title: Intrapulmonary Percussive Ventilation for Children With Bronchiolitis on Non-Invasive Ventilation Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOR-0074-16 CTIL
Record Dates: First submitted 2017-01-29; First posted 2017-01-31 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2016-08

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention)
- Intrapulmonary Percussive Ventilation (Experimental): 15 minutes of IPV physiotherapy
  Interventions: Device: Intrapulmonary Percussive Ventilation (Percussionaire Corp, Sandpoint, Idaho)

INTERVENTIONS:
Device: Intrapulmonary Percussive Ventilation (Percussionaire Corp, Sandpoint, Idaho) — IPV physiotherapy 3 times a day
  Arms: Intrapulmonary Percussive Ventilation

SUMMARY:
Prospective randomized study of patients admitted to the Pediatric Intensive Care Unit suffering from Bronchiolitis and are supported on Non Invasive Positive Pressure Ventilation. The patient population will be divided into two groups, one group will receive conventional treatment and the other group will receive conventional treatment and three times a day of physiotherapy using Intrapulmonary Percussive Ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Bronchiolitis
* PICU patients
* Non Invasive Pressure Support Ventilation
* Age < 24 months

Exclusion Criteria:

* Age > 24 months
* Invasive Ventilation
* No parental consent

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Length of PICU Stay | 10 days
Need for Invasive Ventilation Support | 10 days

SECONDARY OUTCOMES:
S/F ratio | Baseline, 15, 30 and 150 minutes after intervention
  Pulse oximetry saturation/fraction of inspired oxygen
Prevention of lung atelectasis | 10 days
  Per chest x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Cavari, MD, Principal Investigator — Soroka UMC
Locations (1):
- Soroka Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No